CLINICAL TRIAL: NCT04724811
Title: Weight-bearing of Surgically Treated Acetabular Fractures. A Randomised Controlled Trial
Brief Title: Weight-bearing of Surgically Treated Acetabular Fractures.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Kristian Seppänen, Principal Investigator, Hospital District of Helsinki and Uusimaa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/234/2020
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Acetabular Fracture
Keywords: Acetabulum; Periarticular fracture; Weight-bearing
MeSH Terms: interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: Prospective randomised non-inferiority study
Who Masked: Care Provider, Investigator
Masking Description: The surgeon is masked The investigator is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight-bearing as tolerated (Experimental): Patients are instructed to mobilise the hip and weight-bear as tolerated
  Interventions: Procedure: Open reduction and internal fixation (ORIF)
- Touch-down weight-bearing (Active Comparator): Patients are instructed to mobilise the hip. Touch-down weight-bearing for 6-8 weeks
  Interventions: Procedure: Open reduction and internal fixation (ORIF)

INTERVENTIONS:
Procedure: Open reduction and internal fixation (ORIF) — Approaches used:
  * Intrapelvic approach +/- iliac window
  * Kocher-Langenbeck approach

SUMMARY:
The purpose of this study is to determine whether patients with operatively treated acetabular fractures benefit from early weight-bearing as tolerated. The study compares two groups ( n = 25 each), which are randomised into either weight-bearing as tolerated or touch-down weight-bearing for 6-8 weeks postoperatively.

Both study groups are stratified according to

* Type of fracture (anterior approach vs anterior + additional posterior approach)
* Dislocated dome vs non-dislocated/ non existing separate dome fragment

Patients, who are eligible to participate in the trial but choose not to participate in randomisation are asked to enrol in a prospective cohort follow-up cohort. This is to examine a potential participation bias in the RCT groups. These patients will not be counted into the target amount of 50 RCT patients.

DETAILED DESCRIPTION:
For the past 20 years, the established treatment of dislocated acetabular fractures has been surgical reduction and stable osteosynthesis. Good long-term results have been reported in these patients. At present, the mobilisation of these patients after surgery is generally restricted for several weeks ranging from 6-12 weeks touch-down- or non-weight-bearing with no uniform protocol. However there is no scientific evidence for limiting post operative weight-bearing. Accordingly the need of studies on weight-bearing surrounding periarticular fractures has been advocated.

Acetabular fractures in the elderly population are becoming more common and pose significant challenges for treatment including postoperative rehabilitation. Our aim is to investigate if patients benefit of a more liberal weight-bearing regime postoperatively. The primary outcome is measured at 1 year, secondary outcomes are followed up to 10 years postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Unilateral dislocated acetabulum fracture (displacement of over 2mm in preoperative CT scan)
* The osteosynthesis is performed during 21 days after initial trauma
* The patient is willing to participate in the follow-up

Exclusion Criteria:

* Unwillingness to participate in randomisation
* Bilateral fracture
* Letournel & Judet type Both column or Posterior column and wall fractures
* Any other injury that prevents the patient from partial weight bearing
* Open fracture of the acetabulum
* Pathologic fracture (fragility fractures are not an exclusion criteria)
* Prior functional disability in the pelvis or lower extremity
* Non-Compliance due to dementia or other mental disability
* Prior daily pain medication due to hip-pain
* Unwillingness to accept one of the two mobilisation protocols
* Prior hip replacement on injured side
* BMI > 40

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
mHHS | 1 year
  Modified Harris Hip Score, Scale 0-100, higher scores mean better outcome
NRS | 1 year
  Pain during gate, Numerical Rating Scale, Scale 0-10 0=no pain, 10=worst pain

SECONDARY OUTCOMES:
mHHS | 0 weeks, 6 weeks, 12 weeks, 6 months, 2 years, 5 years, 10 years
  Modified Harris Hip Score, Scale 0-100, higher scores mean better outcome
NRS | 0 weeks, 6 weeks, 12 weeks, 6 months, 1 year, 2 years, 5 years, 10 years
  Pain at rest and during gate (2 scores), Numerical Rating Scale, Scale 0-10 0=no pain, 10=worst pain
WOMAC | 0 weeks, 1 year, 2 years, 5 years, 10 years
  Western Ontario and McMaster Universities Osteoarthritis Index, Scale 0-96, higher scores mean better outcome
RAND36 | 0 weeks, 1 Year, 2 years, 5 years, 10 years
  Patient reported quality of life, Scale 0-100, higher scores mean better outcome

OTHER OUTCOMES:
Complications | At any point of time during treatment
  Any complications during treatment are documented
Total hip replacement | During 10 years postoperatively
  Conversion to total hip replacement
Reduction of the articular surface after surgery | Postoperatively
  The reduction is assessed with a postoperative CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Jan Lindahl, MD, PhD, Study Chair — Helsinki University Central Hospital; Kristian Seppänen, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No